CLINICAL TRIAL: NCT00903916
Title: Effect of Weight-increasing Psychotropic Medications on Appetite Regulation
Brief Title: Effect of Antipsychotics on Appetite Regulation
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kimberly Brownley, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: 3024-04003; 1R01MH077117-01A2 (NIH)
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Psychotic Disorders
Keywords: antipsychotic; ghrelin; PYY; appetite; weight gain
MeSH Terms: conditions — Psychotic Disorders; Weight Gain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate changes in appetite-regulating hormones, body composition (weight, body fat%), and hunger ratings in persons early in treatment with one of four atypical antipsychotic medications (olanzapine, risperidone, ziprasidone, aripiprazole).

DETAILED DESCRIPTION:
Severe weight gain and glucose dysregulation are serious problems in patients treated with second-generation ('atypical') antipsychotics (SGA). These side effects frequently interfere with medication compliance and necessitate discontinuation of treatment. Although the causal mechanisms for weight and glucose dysregulation are not well understood, one promising area of investigation targets SGA-induced disturbances in appetite and in appetite-regulating hormones. Findings from our group (and others) demonstrate SGA treatment-related increases in fasting levels of the appetite-stimulating hormone, ghrelin, as well as increases in self-report hunger. This novel study will examine prospective changes in ghrelin and in the 'satiety-signaling' peptide YY (PYY) as measured before and after participants consume a standard mixed-macronutrient meal. Data are obtained at baseline (within 4 weeks of beginning medication), and again 2 months and 4 months later.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM IV criteria for a psychotic disorder (schizophrenia, schizophreniform, brief psychotic disorder, schizoaffective disorder), bipolar disorder, or major depression with psychotic features;
2. "Drug naïve" prior to most recent psychiatric diagnosis;
3. Currently prescribed one of four atypical antipsychotic medications: olanzapine, risperidone, ziprasidone, or aripiprazole;
4. Between the ages of 18 and 40, any race and either gender;
5. Not obese (BMI < 30 kg/m2) (fasting and postprandial ghrelin levels are altered in obesity);
6. Has negative histories for cardiovascular, metabolic, and endocrine disorders at screening;
7. Is willing and able to eat animal-derived foods; and
8. Is not exercising 3 or more times per week.

Exclusion Criteria:

1. Use of medications to treat metabolic and endocrine abnormalities, corticosteroids, over-the-counter appetite suppressants that contain phentermine or Sibutramine;
2. Active involvement with a weight loss program (i.e., Weight Watchers);
3. Serious or unstable medical illness which requires ongoing treatment with medication (this does not include hypertension);
4. Anemia;
5. At serious suicidal risk;
6. Current substance abuse or dependence;
7. For female subjects, pregnancy or nursing (because pregnancy may influence appetite and because the body composition procedure involves low level X-ray exposure).
8. Known history of mental retardation or dementia.
9. Children and adolescents under age 18 will be excluded owing to the inherent confounding effects of normal growth on body weight and appetite.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients ages 18 to 40 years of age who are early in treatment (i.e., started treatment in the past month) with 1 of 4 antipsychotic medications (olanzapine, risperidone, ziprasidone, aripiprazole)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2007-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
ghrelin area under the curve | baseline, 2 and 4 months
PYY area under the curve | baseline, 2 and 4 months

SECONDARY OUTCOMES:
glucose area under the curve | baseline, 2 and 4 months
insulin area under the curve | baseline, 2 and 4 months
body composition | baseline, 2 and 4 months
subjective appetite ratings | baseline, 2 and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Brownley, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Graham KA, Cho H, Brownley KA, Harp JB. Early treatment-related changes in diabetes and cardiovascular disease risk markers in first episode psychosis subjects. Schizophr Res. 2008 Apr;101(1-3):287-94. doi: 10.1016/j.schres.2007.12.476. Epub 2008 Feb 5. PMID 18255275
- [Background] Graham KA, Perkins DO, Edwards LJ, Barrier RC Jr, Lieberman JA, Harp JB. Effect of olanzapine on body composition and energy expenditure in adults with first-episode psychosis. Am J Psychiatry. 2005 Jan;162(1):118-23. doi: 10.1176/appi.ajp.162.1.118. PMID 15625209